CLINICAL TRIAL: NCT05526495
Title: Does a Theory-Based Intervention to Improve Accountability Reduce Low-Value Preoperative Investigations in Patients Undergoing Low Risk Surgery?
Brief Title: Reducing Low-Value Preoperative Investigations in Patients Undergoing Low Risk Surgery
Acronym: Pre-Op
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Jeremy Grimshaw, Senior Scientist, Ottawa Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Reducing Low-Value Pre-Op
Record Dates: First submitted 2022-08-05; First posted 2022-09-02 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Surgery; Anesthesiology
Keywords: Electrocardiographs; Preoperative testing; Chest X-rays; Low Risk Surgical Procedures

STUDY DESIGN:
Intervention Model Description: Eligible hospitals (cluster) within the 26-100th centile for routine preoperative tests will be parallel randomized into two study arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- De-implementation (Experimental): A multi-behaviour technique will be used along with theoretical domains framework.
  Clinicians will be provided with continuing multi-behaviour component intervention to increase accountability for preoperative test ordering in patients having low risk surgeries.
  Interventions: Behavioral: Reducing preoperative low-value test ordering
- Comparator (No Intervention): Standard of care

INTERVENTIONS:
Behavioral: Reducing preoperative low-value test ordering — A multi-component approach will be used:1) An administrative change will be implemented whereby medically necessary preoperative tests for patients undergoing non-urgent surgery will be ordered at the discretion of an anesthesiologist based on their clinical assessment. Adoption of the policy change will be facilitated by a local champion using an engagement and education program for anesthesiologists, surgeons, pre-admission clinic nurses and administrative staff; 2) The workshop program will include rationale for the policy, discussion of perceived local barriers to implementation and mitigation strategies. A train-the-trainer model will be used; 3) The departments will commit to supporting the change in policy. Nurses within preoperative clinic will be coached to feel comfortable calling the anesthesiologist about any pre-op tests ordered, and the Pre-Admission Unit will have the authority to cancel tests that deem unnecessary. Check boxes will be removed from medical order forms
  Arms: De-implementation

SUMMARY:
The purpose of this study is to evaluate if a multi-component behavioral intervention given to anesthesiologists and surgeons is associated with decreasing low value preoperative testing orders in patients undergoing low risk surgery.

The objectives of this trial are to evaluate a) the overall rate of low-value preoperative test (electrocardiogram and chest X-ray) in patients undergoing low risk surgery, b) to conduct an economic and c) process evaluation of the implementation The investigators will assess these outcomes in a sample of 22 Hospitals in Ontario, Canada.

DETAILED DESCRIPTION:
Low-value care is defined as a test or treatment for which there is no evidence of patient benefit or where there is evidence of more harm than benefit.

Within Canada, provincial governments have made reducing low-value care a priority. Choosing Wisely Canada (CWC) is a professionally led campaign that rallies medical professionals to address the issue of low-value care. The CWC makes declarative statements about low-value cares that should be avoided in practice across a broad range of specialties. To date, over 70 Canadian medical specialty societies have developed over 350 recommendations pertaining to unnecessary tests, treatments, and procedures.

Successful de-implementation of low value care require key actors (patients, healthcare providers, managers and policymakers) to change their behaviours and/or decisions while working in complex healthcare environments. Interventions to translate evidence into practice can be effective with the application of behavioural approaches. Behavioural sciences have informed methods for identifying factors that explain and influence behaviour, selecting techniques to address the barriers, and reporting behaviour change interventions. These approaches have yet to be explicitly applied in a systematic and theory-based manner to inform interventions for reducing low-value care.

To address this gap, Grimshaw and colleagues developed the Choosing Wisely De-Implementation Framework (CWDIF), a systematic process framework that uses tools from behavioural science to guide the design, evaluation, and scalability of interventions to reduce low-value care. The CWDIF consists of five phases: Phase 0, identification of potential areas of low-value healthcare; Phase 1, identification of local priorities for implementation of CWC recommendations (i.e., de-implementing low-value care); Phase 2, identification of barriers to implementing CWC recommendations and potential interventions to overcome these; Phase 3, rigorous evaluations of CWC implementation programmes; and Phase 4, spread of effective CWC implementation programmes.

In Canada, CWC provides a list of items that are considered low-value care for each medical specialty and provincial CWC campaigns have prioritized the items that are relevant to each province (Phase 0). The Canadian Anesthesiologists Society made 3 CWC recommendations against routine pre-operative tests prior to low risk surgery. In 2015, CWC and Health Quality Ontario co-hosted a stakeholder event of 60 key health system leaders in Ontario who identified low value preoperative testing, such as electrocardiographs and chest X-rays prior to low risk surgery as a key priority (Phase 1). Having identified the local priorities, it is important to identify determinants (barriers and enablers) of the particular low-value care that can be address by intervention (Phase 2). A theory-based qualitative study with Ontario anesthesiologists and surgeons used the Theoretical Domains Framework to understand individual, socio-cultural, and environmental factors that influence behaviour in specific contexts. Barriers identified included conflict about who was responsible for the test-ordering (Social/professional role and identity), inability to cancel tests ordered by fellow physicians (Beliefs about capabilities and Social influences), and logistic problems with tests being completed before the anesthesiologists see the patient (Beliefs about capabilities and Environmental context and resources). There were also concerns that not testing might be associated with harms (Beliefs about Consequences). These findings led to the development of a theory-informed intervention that identifies anesthesiologists as the primary focus for ordering of tests and strengthens accountability within hospitals.

The next phase of the framework requires the evaluation of the theory-informed intervention (Phase 3).This study is a cluster randomized controlled trial in 22 hospitals in Ontario, Canada to determine if preoperative testing ordered by anesthesiologist and supported by a focused implementation strategy can decrease the use of low-value preoperative tests in patients undergoing low risk surgeries.

ELIGIBILITY:
The study intervention will target hospitals, anesthesiologists, surgeons, pre-admission clinic nurses, and administrative staff.

Cluster (Hospital) Level Inclusion Criterion:

1. Hospitals in Ontario, Canada
2. within the 26-100th centile for routine preoperative tests for 2019

The study will recruit anesthesiologist and surgeons taking care of patients that meet the following criterion:

Patient Level Inclusion Criterion:

1. ≥18 age
2. undergoing low risk surgeries such as:

   * endoscopy
   * ophthalmologic surgery
   * knee arthroscopy
   * hernia repair

Exclusion Criteria:

* emergency elective chest X-rays and/or electrocardiogram

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Pre-operative testing | within 60 days before surgery
  Proportion of patients receiving one or more low-value preoperative tests within 60 days before surgery

SECONDARY OUTCOMES:
Overnight admission | within 24 hours from the date of surgery
  proportions of patients with overnight admission
Re-operation events | within 24 hours
  rate of re-operation within 24 hours after primary surgery
All-cause mortality | 30-day from the date of surgery
  30-day all-cause mortality from the date of surgery
Preoperative tests | 6 months
  proportions of patients receiving each of the included preoperative investigations individually
Mechanistic sub-study | 6 months
  We will test whether changes in healthcare providers' behaviour are mediated through changes in hypothesized mechanisms using bootstrapped multiple mediation models controlling for hospital clustering and baseline response
Economic Evaluation | 6 months
  We will compare the total costs of the intervention to the total costs of the control group. Results will be presented as an incremental cost per one preoperative test avoided. The monetary cost will be estimated using micro-costing technique by measuring monetary costs associated with perioperative assessment, hospital admissions and re-operations will be derived from ICES databases, and patient out-of-pocket costs and time missed from work because of attending pre-op tests such as chest x-rays and echocardiographs
Fidelity evaluation | 1 month
  In the intervention arm only we will conduct a fidelity check-intervention checklist to assess: low; medium; high risk, with a semi-structured interview with physicians in the intervention arm. De-identified interviews will be analyzed by two independent researchers using the content analysis. A descriptive analysis will be used to summarize all data and a fidelity score will be calculated from a 7 point Likert scale (1:strongly agree; 7: strongly disagree).

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Grimshaw, PhD, Study Director — Ottawa Hospital Research Institute; Kyle Kirkham, MD, Principal Investigator — Department of Anaesthesia, Toronto Western Hospital, University of Toronto
Locations (4):
- Canada (4):
  - Muskoka Algonquin Healthcare, Muskoka, Onario
  - Grand River Hospital, Kitchener, Ontario
  - St.Joseph'S Health Care, London, Ontario
  - Stratford General Hospital, Stratford, Ontario

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available at the moment. Aggregated cluster level data may be share upon reasonable request once the study has been published.

REFERENCES:
- [Background] Grimshaw JM, Patey AM, Kirkham KR, Hall A, Dowling SK, Rodondi N, Ellen M, Kool T, van Dulmen SA, Kerr EA, Linklater S, Levinson W, Bhatia RS. De-implementing wisely: developing the evidence base to reduce low-value care. BMJ Qual Saf. 2020 May;29(5):409-417. doi: 10.1136/bmjqs-2019-010060. Epub 2020 Feb 6. PMID 32029572
- [Background] Kirkham KR, Wijeysundera DN, Pendrith C, Ng R, Tu JV, Laupacis A, Schull MJ, Levinson W, Bhatia RS. Preoperative testing before low-risk surgical procedures. CMAJ. 2015 Aug 11;187(11):E349-E358. doi: 10.1503/cmaj.150174. Epub 2015 Jun 1. PMID 26032314
- [Background] Patey AM, Islam R, Francis JJ, Bryson GL, Grimshaw JM; Canada PRIME Plus Team. Anesthesiologists' and surgeons' perceptions about routine pre-operative testing in low-risk patients: application of the Theoretical Domains Framework (TDF) to identify factors that influence physicians' decisions to order pre-operative tests. Implement Sci. 2012 Jun 9;7:52. doi: 10.1186/1748-5908-7-52. PMID 22682612